CLINICAL TRIAL: NCT01232374
Title: A Clinical Study of Nimotuzumab in Combination With Concurrent Chemotherapy and Radiation for Patients With Local Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Nimotuzumab in Combination With Chemoradiation for Local Advanced Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BT-ESO-1001
Record Dates: First submitted 2010-10-12; First posted 2010-11-02 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Squamous Cell Carcinoma
Keywords: Nimotuzumab; local advanced esophageal squamous cell carcinoma; chemo-irradiation
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — nimotuzumab; Cisplatin; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nimotuzumab plus chemo-irradiation (Experimental): Nimotuzumab，chemotherapy(cisplatin )，radiotherapy
  Interventions: Drug: Nimotuzumab; Drug: cisplatin; Radiation: Radiotherapy
- Placebo plus chemo-irradiation (Placebo Comparator): Placebo，chemotherapy(cisplatin)，radiotherapy
  Interventions: Drug: Placebo; Drug: cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Nimotuzumab — 200mg (4 bottles), once a week for 7 weeks during irradiation (week 1, week 2, week 3, week 4, week 5, week 6 and week 7). After irradiation 200mg (4 bottles), once every 4 weeks for 2 cycles (week 9 and week 13)
  Arms: Nimotuzumab plus chemo-irradiation
Drug: Placebo — 4 bottles placebo, once a week for 7 weeks during irradiation (week 1, week 2, week 3, week 4, week 5, week 6 and week 7). After irradiation 200mg (4 bottles), once every 4 weeks for 2 cycles (week 9 and week 13)
  Other Names: Nimotuzumab, Placebo
  Arms: Placebo plus chemo-irradiation
Drug: cisplatin — cisplatin 25 mg/m2/d, d1-3, once every 4 weeks for 4 cycles (week 1, week 5, week 9 and week 13); 5-FU 600 mg/m2/d, d1-3, continuously infusion for 72 hrs,once every 4 weeks for 4 cycles (week 1, week 5, week 9 and week 13).
Radiation: Radiotherapy — A total dose of 61.2 Gy will be delivered in 34 fractions at 1.8 Gy/fraction, 5 fractions per week in 6.8 weeks.
  Placebo: 4 bottles placebo, once a week for 7 weeks during irradiation (week 1, week 2, week 3, week 4, week 5, week 6 and week 7). After irradiation 200mg (4 bottles), once every 4 weeks for 2 cycles (week 9 and week 13)

SUMMARY:
Nimotuzumab is a humanized monoclonal antibody against epidermal growth factor receptor (EGFR). Clinical trials are ongoing globally to evaluate Nimotuzumab in different indications. Nimotuzumab has been approved to treat squamous cell carcinoma of head and neck (SCCHN), glioma and nasopharyngeal carcinoma in different countries. The clinical phase I study of the combination of Nimotuzumab administered concurrently with chemo-irradiation in patients with local advanced esophageal squamous cell carcinoma (LAFSCC) has shown the safety and the potential efficacy of Nimotuzumab. The concurrent trial is a clinical phase II trial designed to assess the efficacy of the combination of Nimotuzumab administered concurrently with chemo-radiotherapy in patients with LAFSCC, and to further investigate its side-effect and toxicity.

DETAILED DESCRIPTION:
The concurrent trial is a clinical phase II trial designed to assess the efficacy of the combination of Nimotuzumab administered concurrently with chemo-radiotherapy in patients with LAFSCC, and to further investigate its side-effect and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Joined the study voluntarily and signed informed consent form;
* Age 18-75
* Both genders
* Esophageal squamous cell carcinoma confirmed by pathology
* Local advanced esophageal squamous cell carcinoma (T2N0M0-TxNxM1a, AJCC 2002)
* No radiotherapy, chemotherapy or other treatments prior to enrollment
* PS ECOG 0-2
* Life expectancy of more than 3 months
* Target lesions measurable
* Hemoglobin（Hb）≥9 g/dL
* WBC≥3x109/L, Neutrophils (ANC )≥1.5x109/L
* platelet count (Pt) ≥100x 109/L
* Hepatic function: ALAT and ASAT < 2.5 x ULN, TBIL<1.5 x ULN
* Renal function: creatinine < 1.5 x ULN
* No immuno-deficiency
* Use of an effective contraceptive for adults to prevent pregnancy.

Exclusion Criteria:

* Complete esophageal obstruction
* Deep esophageal ulcer
* Esophageal perforation
* Haematemesis
* After surgery, exploratory thoracotomy, radiotherapy, chemotherapy, or targeting therapy
* Esophageal stent or tracheal stent placed
* Other malignant tumors, except for skin basal cell carcinoma, or cervical carcinoma in situ, who survived with no evidence disease for over 3 years
* Participation in other interventional clinical trials within 30 days
* Pregnant or breast-feeding women or people during the birth-period who refused to take contraceptives
* Drug addiction
* Alcoholism or AIDS
* Uncontrolled seizures or psychiatric diseases, loss of control over their own behavior
* History of serious allergic or allergy
* Patients who are not suitable to participate in the trial according to researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2010-09; Primary Completion 2015-10 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Response rate of Nimotuzumab combined with chemo-irradiation | 2 months after radiotherapy
1-yr overall survivals | 1 year
2-yr overall survival | 2 year
3-yr overall survival | 3 years

SECONDARY OUTCOMES:
Local progression-free survival | 3 years
Disease progression-free survival | 3 years
Distant metastasis rate | 3 years
Number and grade of Participants with Adverse Events | 6 months
Quality of life | 3 years

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Chinese Academy of Medical Sciences Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Provincial Tumor Hospital, Fuzhou, Fujian
  - Cancer Center of Sun Yat-sen, Guangzhou, Guangdong
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Huazhong University of Science and Technology, Union Hospital, Tongji Medical College, Wuhan, Hubei
  - Cancer Hospital of Jiangsu Province, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University,Suzhou First People's Hospital, Suzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The first bethune hospital of Jilin university, Changchun, Jilin
  - Affiliated Hospital of Qingdao University Medical College, Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Fourth Military Medical University Xijing Hospital, Xian, Shanxi
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang